CLINICAL TRIAL: NCT06577987
Title: A Phase 1, Open-Label, Multicenter Study to Evaluate the Safety and Efficacy of the Oral Cyclin A/B-RxL Inhibitor CID-078 in Patients With Advanced Solid Tumor Malignancies
Brief Title: Safety/Efficacy Study of CID-078 in Patients With Advanced Solid Tumor Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Circle Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CID-AB1-24001
Record Dates: First submitted 2024-08-23; First posted 2024-08-29 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-05

CONDITIONS: Advanced Solid Tumor; Metastatic Solid Tumor; Refractory Solid Tumor; Cancer; Lung Cancer; Triple Negative Breast Cancer; Breast Neoplasms; Neuroendocrine Tumors; Neuroendocrine Carcinoma; RB1 Gene Mutation
Keywords: Phase 1; CID-078; Estrogen
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms; Lung Neoplasms; Triple Negative Breast Neoplasms; Breast Neoplasms; Neuroendocrine Tumors; Carcinoma, Neuroendocrine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Part 1a Dose Escalation, Part 1b New Formulation/Pilot Food Effect and Part 2 Dose Expansion (Experimental)
  Interventions: Drug: CID-078 Monotherapy

INTERVENTIONS:
Drug: CID-078 Monotherapy — Cyclin A/B-RxL inhibitor, twice-a-day in repeating 21-day treatment cycles until disease progression or discontinuation criteria.

SUMMARY:
This is a first-in-human, multicenter, open-label, phase 1 study to evaluate safety, tolerability, and efficacy of CID-078, a Cyclin A/B-RxL inhibitor, in patients with advanced solid tumors.

DETAILED DESCRIPTION:
This is a first-in-human, multicenter, open-label, phase 1 study to evaluate safety, tolerability, and efficacy of CID-078, a Cyclin A/B-RxL (Arginine-any amino acid-lysine) inhibitor, in patients with advanced solid tumors. The study will be conducted at approximately 20 centers. CID-078 will be evaluated as an oral therapeutic. This study is divided into three parts: Part 1a Dose Escalation, Part 1b New Formulation Dose Escalation/Pilot Food Effect and Part 2 Dose Expansion.

Part 1a will evaluate safety, tolerability, pharmacokinetics and pharmacodynamics of CID-078, and identify recommended dose for expansion (RDE) of CID-078 using a Backfill Bayesian Optimal Interval design. Dose escalation will occur sequentially over several dose levels.

Part 1b will evaluate the safety and tolerability of a new CID-078 oral formulation, investigate the pharmacokinetic exposure between the original and new CID-078 formulations, and evaluate the effect of food on CID-078 pharmacokinetics. Part 1b will be initiated upon availability of the new CID-078 oral formulation.

Part 2 is a Dose Expansion. Upon identification of the RDE as determined by the SRC, CID-078 will be further evaluated for it's antitumor activity/efficacy along with characterization of it's safety, tolerability, pharmacokinetics, and pharmacodynamics in three tumor specific cohorts: TNBC, SCLC, and solid tumors harboring a RB1 alteration or Rb protein LoF; with an additional possible cohort expansion of N=20 for either TNBC or RB1-altered solid tumor cohort based on data observed.

The study consists of a 28-day Screening Period, a Treatment Period, an End of Treatment (EOT) Visit, and a Safety Follow-up Visit. After confirming eligibility, patients enter the Treatment Period that consists of repeating 21-day treatment cycles. Study drug treatment cycles will continue for as long as the patient does not meet study drug discontinuation criteria. Within 7 days of the last dose of study drug or the decision to withdraw from the study, patients will undergo an EOT visit and a Safety Follow-Up visit 28 days after the EOT visit.

ELIGIBILITY:
Part 1a/1b Inclusion Criteria:

A patient must meet all of the following inclusion criteria to be eligible to participate in this study.

1. Solid tumor malignancy meeting the following criteria:

   * Part 1a Dose Escalation and Part 1b New Formulation Dose Escalation/Pilot Food Effect Cohort: locally advanced or metastatic solid tumor malignancy that has progressed or was non responsive to available therapies and for which no standard or available curative therapy exists.
   * Part 1a and Part 1b Backfill: patients with TNBC, SCLC, and solid tumors harboring a RB1 or CDKN2A/B loss genomic alteration or Rb protein LoF. Additional tumor types or genomic alterations may be considered by the SRC as data become available. Patient must have progressed or was non-responsive to available therapies and for which no standard or available curative therapy exists
2. Measurable disease per RECIST v1.1.
3. Age ≥ 18 years.
4. Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
5. Life expectancy > 12 weeks.
6. Able to undergo a fresh biopsy if medically feasible.
7. Ability to swallow capsules by mouth.
8. Have the following laboratory values:

   1. Calculated creatinine clearance (CrCl) ≥ 60 mL/min/1.73 m^2 by Cockroft-Gault formula (actual body weight must be used for CrCl unless body mass index [BMI] is > 30 kg/m2, then lean or ideal body weight must be used (based on institutional practice), or estimated glomerular filtration rate (eGFR) ≥ 60 mL/min/1.73 m2 based alternative methods of determination (e.g., modification of diet in renal disease [MDRD], 24-hour urine collection) if consistent with local or institutional practice.
   2. Total bilirubin ≤ 1.5 × upper limit of normal (ULN) unless prior history of Gilbert's syndrome with Sponsor Medical Monitor approval.
   3. Aspartate transaminase and alanine transaminase ≤ 2.5 × ULN, or ≤ 5 × ULN if due to liver involvement by tumor.
   4. Hemoglobin ≥ 9.0 g/dL (last transfusion > 14 days prior to first dose of study drug).
   5. Platelets ≥ 100 × 10^9 cells/L (last platelet transfusion > 14 days prior to first dose of study drug).
   6. Absolute neutrophil count ≥ 1.2 × 10^9 cells/L (last dose of hematopoietic growth factors > 14 days from first dose of study drug).
9. Females of childbearing potential must commit to sexual abstinence or to use two acceptable forms of birth control (defined as the use of an intrauterine device, a barrier method with spermicide, condoms, or any form of hormonal contraceptives) for the duration of the study and for four months following the last dose of study treatment. Females who are at least two years postmenopausal or premenopausal with documented hysterectomy, bilateral salpingectomy, bilateral oophorectomy, or permanent infertility due to alternate medical causes other than above are not considered females of childbearing potential. Male patients must be sterile (biologically or surgically), commit to sexual abstinence or to the use of a reliable method of birth control (condoms with spermicide) for the duration of the study and for four months following the last dose of study treatment.
10. Females of childbearing potential must have a negative serum pregnancy test during Screening and a negative urine or serum pregnancy test prior to receiving the first dose of study drug. Females who are at least two years postmenopausal or premenopausal with documented hysterectomy, bilateral salpingectomy, bilateral oophorectomy, or permanent infertility due to alternate medical causes other than above are not considered females of childbearing potential.
11. Signed and dated Institutional Review Board (IRB)/Ethics Committee (EC)-approved ICF before any protocol-directed screening procedures are performed.

    Part 1b Pilot Food Effect Cohort - Specific Inclusion Criteria

    Patients who consent to participate in the pilot food effect cohort will also be required to meet the following inclusion criteria:
12. Able to eat a standardized high-fat, high-caloric or low-fat meal (as applicable to the food effect cohort assigned) within 25 minutes.

Exclusion Criteria:

A patient who meets any of the following exclusion criteria will be ineligible to participate in this study:

1. Treatment with any of the following:

   1. Targeted therapy ≤ eight days or 5× the terminal phase elimination half-lives, whichever is shorter, prior to the first dose of study drug.
   2. Systemic anticancer treatment (excluding targeted therapy as described above) ≤ 14 days prior to first dose of study drug.
   3. Radiotherapy ≤ 28 days and palliative radiation ≤ 14 days prior to the first dose of study drug. If irradiated, lesions must have demonstrated clear-cut progression prior to being eligible for evaluation as target lesions.
   4. Immunotherapy ≤ 28 days prior to the first dose of study drug.
   5. Major surgery ≤ 28 days prior to the first dose of study drug.
2. Have any unresolved toxicity of Grade ≥ 2 from previous anti-cancer treatment, except for alopecia and skin pigmentation. Patients with chronic, but stable Grade 2 toxicities may be allowed to enroll after agreement between the Investigator and Sponsor Medical Monitor.
3. Have known or suspected brain metastases or spinal cord compression, unless the condition has been asymptomatic, treated with surgery and/or radiation, and has been stable without requiring escalating doses of corticosteroids or anti-convulsant medications for at least four weeks prior for the first dose of study drug.
4. Prior therapy with CID-078.
5. Known hypersensitivity to CID-078 or any drugs similar in structure or class.
6. Past medical history of interstitial lung disease, or any evidence of clinically active interstitial lung disease. Patients with sub-clinical pneumonitis who have received anti-cancer therapy (e.g., immunotherapy, ADC) previously can be included if their condition is stable without any medical intervention.
7. Patient has a history of congestive heart failure (CHF) Class III/IV according to the New York Heart Association (NYHA) Functional Classification or serious cardiac arrhythmias requiring treatment.
8. Heart rate corrected QT (QTc) interval (using Fridericia correction calculation) > 470 msec.
9. Current treatment with medication known to prolong the QT/QTc interval (see examples from Table 28) or history of additional risk factors for Torsade de Pointes (e.g., heart failure, Grade ≥ 3 hypokalemia, family history of long QT syndrome). Patient who has adequately controlled condition or requires use of medications from Table 28 may be allowed upon agreement by the Investigator and Sponsor Medical Monitor.
10. Pregnant or lactating women.
11. History of another primary malignancy ≤ two years prior to starting study drug, except for adequately treated cancer (e.g., basal, or squamous cell carcinoma of the skin or cancer of the cervix in situ).
12. Malabsorption syndrome or other conditions (e.g., refractory nausea and vomiting, external biliary diversion, or any significant small bowel resection) that may interfere with adequate absorption of investigational product.
13. Uncontrolled intercurrent illness including, but not limited to, uncompensated respiratory, cardiac, hepatic, or renal disease, active infection (including untreated human immunodeficiency virus [HIV] and active clinical tuberculosis), symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
14. Current endocrinopathies, unless in the opinion of the Investigator, endocrine complications are stable and well controlled and study participation does not jeopardize patient's health and wellbeing. Patients with asymptomatic endocrine disease on endocrine replacement therapy are eligible.
15. Active hepatitis B infection as defined by a positive hepatitis B surface antigen (HbsAg) test and detectable hepatitis B virus (HBV) DNA. Patients ineligible due to detectable levels of HBV DNA at baseline may be rescreened for enrollment if their HBV DNA levels become undetectable after treatment with antiviral agents, and upon agreement between the Investigator and Sponsor Medical Monitor.
16. Active hepatitis C infection as defined by a reactive hepatitis C virus (HCV) antibody test and detectable HCV RNA.
17. For patients with a history of HIV or acquired immunodeficiency syndrome (AIDS):

    1. Must have a CD4+ T-cell count ≥ 350 cells/μL
    2. Have not had an opportunistic infection within the previous 12 months.
    3. To be on current antiretroviral therapy (ART) regimen for a minimum of four weeks and have an HIV viral load < 400 copies/mL at the time of enrollment.
    4. Patients who are using concurrent strong cytochrome P450 (CYP)3A4 inhibitors (e.g., ritonavir, cobicistat) or strong CYP3A4 inducers are excluded from the study if their regimen cannot be altered. Otherwise, eligible study patients could be switched to an alternate effective ART before study participation.
18. Current treatment with a strong CYP3A4 inhibitor or inducer, Pgp inhibitor, or CYP3A4 sensitive substrate within 14 days or five terminal half-lives prior to the first dose of study drug, whichever is shorter.
19. Active bleeding disorders.
20. Prior solid organ transplantation.
21. Is, in the Investigator's opinion, unable or unwilling to comply with the study procedures.
22. Have any condition or illness that, in the opinion of the Investigator, might compromise patient safety or interfere with the evaluation of the safety of the study drug.

Study Population (Part 2 Dose Expansion):

Inclusion Criteria:

A patient must meet all of the following inclusion criteria to be eligible to participate in this study.

1. Advanced or metastatic solid tumor malignancy that has progressed or was non responsive to available therapies and for which no standard or available curative therapy exists.

   1. Triple negative breast cancer (TNBC) cohort: histologically or cytologically confirmed TNBC per American Society for Clinical Oncology/College of American Pathologists (ASCO/CAP) criteria, based on the most recent analyzed biopsy or other pathology specimen.
   2. Small cell lung cancer (SCLC) cohort: histologically or cytologically confirmed relapsed/refractory SCLC.
   3. Retinoblastoma 1 (RB1)-altered solid tumor cohort: solid tumors harboring a documented RB1 genomic alteration or Rb protein LoF, as identified through assays performed at Clinical Laboratory Improvement Amendments (CLIA)-certified or other similarly certified laboratories.
2. Patients must have measurable disease by RECIST v1.1.
3. Age ≥ 12 years and at least 40 kg in body weight.
4. Eastern Cooperative Oncology Group (ECOG) performance status 0-1 (patients ≥ 18 years of age), Karnofsky performance status ≥ 70% (patients ≥ 16 to < 18 years of age), or Lansky performance status ≥ 70% (patients < 16 years of age). Patients who are unable to walk because of paralysis, but who can sit in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score (Appendix 1).
5. Life expectancy >12 weeks.
6. For patients ≥ 18 years of age: able to undergo a fresh biopsy if medically feasible.
7. Ability to swallow capsules by mouth.
8. Have the following laboratory values:

   1. For patients ≥ 18 years of age: calculated CrCl ≥ 60 mL/min/1.73 m2 by Cockroft-Gault formula (actual body weight must be used for CrCl unless BMI > 30 kg/m2 then lean or ideal body weight must be used based on institutional practice), or estimated glomerular filtration rate (eGFR) ≥ 60 mL/min/1.73 m2 based alternative methods of determination (e.g., modification of diet in renal disease [MDRD], 24-hour urine collection) if consistent with local or institutional practice. For patients < 18 years of age: serum creatinine within normal limits (as defined below) or estimated glomerular filtration rate (eGFR) ≥ 60 mL/min/1.73 m2 based on local institutional practice for determination.

      Age at Screening Maximum Serum Creatinine SI Unit age 12 to < 15 years - 0.81 mg/dL; age 15 to < 18 years (male) - 1.08 mg/dL; age 15 to < 18 years (female) - 0.84 mg/dL
   2. Total bilirubin ≤ 1.5 × ULN unless prior history of Gilbert's syndrome with Sponsor Medical Monitor approval.
   3. Aspartate transaminase and alanine transaminase ≤ 2.5 × ULN, or ≤ 5 × ULN if due to liver involvement by tumor.
   4. Hemoglobin ≥ 9.0 g/dL (last transfusion > 14 days prior to first dose of study drug).
   5. Platelets ≥ 100 × 10^9 cells/L (last platelet transfusion > 14 days prior to first dose of study drug).
   6. Absolute neutrophil count ≥ 1.2 ×10^9 cells/L (last dose of hematopoietic growth factors > 14 days from first dose of study drug).
9. Females of childbearing potential must commit to sexual abstinence or to use two acceptable forms of birth control (defined as the use of an intrauterine device, a barrier method with spermicide, condoms, any form of hormonal contraceptives) for the duration of the study and for four months following the last dose of study treatment. Females who are at least two years postmenopausal or premenopausal with documented hysterectomy, bilateral salpingectomy, bilateral oophorectomy, or permanent infertility due to alternate medical causes other than above are not considered females of childbearing potential. Male patients must be sterile (biologically or surgically), commit to sexual abstinence or to the use of a reliable method of birth control (condoms with spermicide) for the duration of the study and for four months following the last dose of study treatment.
10. Females of childbearing potential must have a negative serum pregnancy test during Screening and a negative urine or serum test prior to receiving first dose of study drug. Females who are at least two years postmenopausal or premenopausal with documented hysterectomy, bilateral salpingectomy, bilateral oophorectomy, or permanent infertility due to alternate medical causes other than above are not considered females of childbearing potential.
11. Signed and dated IRB/EC-approved ICF for potential patients ≥ 18 years of age. A signed and dated IRB/EC-approved adolescent assent form may also be required for patients 12 to 17 years of age in addition to an ICF signed by a parent or legal guardian.

Exclusion Criteria:

A patient who meets any of the following exclusion criteria will be ineligible to participate in this study.

1. Treatment with any of the following:

   1. Targeted therapy ≤ eight days or 5× the terminal phase elimination half-lives, whichever is shorter, prior to the first dose of study drug.
   2. Systemic anticancer treatment (excluding targeted therapy as described above) ≤ 14 days prior to the first dose of study drug.
   3. Radiotherapy ≤ 28 days and palliative radiation ≤ 14 days prior to the first dose of study drug. If irradiated, lesions must have demonstrated clear-cut progression prior to being eligible for evaluation as target lesions.
   4. Immunotherapy ≤ 28 days prior to the first dose of study drug.
   5. Major surgery ≤ 28 days prior to the first dose of study drug.
2. Have any unresolved toxicity of Grade ≥ 2 from previous anti-cancer treatment, except for alopecia and skin pigmentation. Patients with chronic, but stable Grade 2 toxicities may be allowed to enroll after agreement between the Investigator and Sponsor Medical Monitor.
3. Have known or suspected brain metastases or spinal cord compression, unless the condition has been asymptomatic, treated with surgery and/or radiation, and has been stable without requiring escalating doses of corticosteroids or anti-convulsant medications for at least four weeks prior to the first dose of study drug.
4. Prior therapy with CID-078.
5. Known hypersensitivity to CID-078 or any drugs similar in structure or class.
6. Past medical history of interstitial lung disease or any evidence of clinically active interstitial lung disease. Patients with sub-clinical pneumonitis who have received anti-cancer therapy (e.g., immunotherapy, ADC) previously can be included if their condition is stable without any medical intervention.
7. Patient has a history of CHF Class III/IV according to the NYHA Functional Classification Appendix 2) or serious cardiac arrhythmias requiring treatment.
8. QTc interval (using Fridericia correction calculation) (QTcF) > 470 msec.
9. Current treatment with medication known to prolong the QT/QTcF interval or history of additional risk factors for Torsade de Pointes (e.g., heart failure, Grade ≥ 3 hypokalemia, family history of long QT syndrome). Patient who has adequately controlled condition or require use of medications from Table 28 may be allowed to enroll upon agreement by the Investigator and Sponsor Medical Monitor.
10. Pregnant or lactating women.
11. History of another primary malignancy ≤ two years prior to starting study drug, except for adequately treated cancer (e.g., basal or squamous cell carcinoma of the skin or cancer of the cervix in situ).
12. Malabsorption syndrome or other conditions (e.g., refractory nausea and vomiting, external biliary diversion, or any significant small bowel resection) that may interfere with adequate absorption of investigational product.
13. Uncontrolled intercurrent illness including, but not limited to, uncompensated respiratory, cardiac, hepatic, or renal disease, active infection (including untreated HIV and active clinical tuberculosis), symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
14. Current endocrinopathies, unless in the opinion of the Investigator, endocrine complications are stable and well controlled and study participation does not jeopardize patient's health and wellbeing. Patients with asymptomatic endocrine disease on endocrine replacement therapy are eligible.
15. Active hepatitis B infection as defined by a positive HBsAg test and detectable HBV DNA. Patients ineligible due to detectable levels of HBV DNA at baseline may be rescreened for enrollment if their HBV DNA levels become undetectable after treatment with antiviral agents, and upon agreement between the Investigator and Sponsor Medical Monitor.
16. Active hepatitis C infection as defined by a reactive HCV antibody test and detectable HCV RNA.
17. For patients with a history of HIV or AIDS:

    1. Must have a CD4+ T-cell count ≥ 350 cells/μL.
    2. Have not had an opportunistic infection within the previous 12 months.
    3. To be on current ART regimen for a minimum of four weeks and have an HIV viral load < 400 copies/mL at the time of enrollment.
    4. Patients who are using concurrent strong CYP3A4 inhibitors (e.g., ritonavir, cobicistat) or strong CYP3A4 inducers are excluded from the study if their regimen cannot be altered. Otherwise, eligible study patients could be switched to an alternate effective ART regimen before study participation.
18. Current treatment with a strong CYP3A4 inhibitor or inducer, Pgp inhibitor, or CYP3A4 sensitive substrate as specifically listed in Table 26 and Table 27 within 14 days or five terminal half-lives prior to the first dose of study drug, whichever is shorter.
19. Active bleeding disorders.
20. Prior solid organ transplantation.
21. Is, in the Investigator's opinion, unable or unwilling to comply with the study procedures.
22. Have any condition or illness that, in the opinion of the Investigator, might compromise patient safety or interfere with the evaluation of the safety of the study drug.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2024-08-14 (Actual); Primary Completion 2027-01-14 (Estimated); Study Completion 2027-03-14 (Estimated)

PRIMARY OUTCOMES:
Part 1: Incidence of Treatment Emergent Adverse Events (TEAEs) based on CTCAE v5.0. | From first dose of CID-078 on Cycle 0 Day 1/ Cycle 1 Day 1 (each cycle is 21 days) to 28 days after the last dose of study drug.
Part 1: Incidence of Treatment Related Adverse Events (TRAEs) based on CTCAE v5.0. | From first dose of CID-078 on Cycle 0 Day 1/ Cycle 1 Day 1 (each cycle is 21 days) to 28 days after the last dose of study drug.
Part 1: Incidence of Dose-Limiting Toxicities (DLTs). | From first dose of CID-078 on Cycle 0 Day 1/ Cycle 1 Day 1 (each cycle is 21 days) to end of cycle 1, up to 21 + 4 days.
Part 1: To determine recommended dose(s) for expansion (RDEs) for evaluation for Part 2. | From first dose of CID-078 on Cycle 0 Day 1/ Cycle 1 Day 1 (each cycle is 21 days) to 28 days after the last dose of study drug.
  The RDEs will be determined using all available information, including, but not limited to, AEs, dose-limiting toxicities, pharmacokinetic parameters, clinical laboratory tests, and efficacy measures observed in Part 1 Dose Escalation.
Part 2: Percentage of patients with confirmed objective response per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 Criteria in Solid Tumors. | From first dose of CID-078 on Cycle 0 Day 1/ Cycle 1 Day 1 (each cycle is 21 days) to 28 days after the last dose of study drug.
Part 2: Duration of confirmed objective response per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 Criteria in Solid Tumors. | From first dose of CID-078 on Cycle 0 Day 1/ Cycle 1 Day 1 (each cycle is 21 days) to 28 days after the last dose of study drug.
Part 2: Duration of disease progression free survival per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 Criteria in Solid Tumors. | From first dose of CID-078 on Cycle 0 Day 1/ Cycle 1 Day 1 (each cycle is 21 days) to 28 days after the last dose of study drug.
Part 2: To determine Provisional Recommended Phase 2 Dose (RP2D) for future dose optimization. | From first dose of CID-078 on Cycle 0 Day 1/ Cycle 1 Day 1 (each cycle is 21 days) to 28 days after the last dose of study drug.
  Provisional RP2D will be determined using all available information, including, but not limited to, Adverse Events (AEs), dose-limiting toxicities, pharmacokinetic parameters, clinical laboratory tests, and efficacy measures observed during the study.

SECONDARY OUTCOMES:
Part 1: Percentage of patients with confirmed objective response per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 Criteria in Solid Tumors. | From first dose of CID-078 on Cycle 0 Day 1/ Cycle 1 Day 1 (each cycle is 21 days) to 28 days after the last dose of study drug.
Part 1: Duration of confirmed objective response per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 Criteria in Solid Tumors. | From first dose of CID-078 on Cycle 0 Day 1/ Cycle 1 Day 1 (each cycle is 21 days) to 28 days after the last dose of study drug.
Part 1: Duration of disease progression free survival per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 Criteria in Solid Tumors. | From first dose of CID-078 on Cycle 0 Day 1/ Cycle 1 Day 1 (each cycle is 21 days) to 28 days after the last dose of study drug.
Part 1: Maximum plasma concentration (Cmax) of CID-078 in fasted and fed state. | From first dose of CID-078 on Cycle 0 Day 1/ Cycle 1 Day 1 (each cycle is 21 days) to 28 days after the last dose of study drug.
Part 1: Time to maximum plasma concentration (Tmax) of CID-078 in fasted and fed state. | From first dose of CID-078 on Cycle 0 Day 1/ Cycle 1 Day 1 (each cycle is 21 days) to 28 days after the last dose of study drug.
Part 1: Area under the concentration-time curve (AUC) of CID-078 in fasted and fed state. | From first dose of CID-078 on Cycle 0 Day 1/ Cycle 1 Day 1 (each cycle is 21 days) to 28 days after the last dose of study drug.
Part 1 and Part 2: Terminal half-life (t1/2) of CID-078 in fasted and fed state. | From first dose of CID-078 on Cycle 0 Day 1/ Cycle 1 Day 1 (each cycle is 21 days) to 28 days after the last dose of study drug.
Part 2: Incidence of Treatment Emergent Adverse Events (TEAEs) based on CTCAE v5.0. | From first dose of CID-078 on Cycle 0 Day 1/ Cycle 1 Day 1 (each cycle is 21 days) to 28 days after the last dose of study drug.
Part 2: Incidence of Treatment Related Adverse Events (TRAEs) based on CTCAE v5.0. | From first dose of CID-078 on Cycle 0 Day 1/ Cycle 1 Day 1 (each cycle is 21 days) to 28 days after the last dose of study drug.

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Florida Cancer Specialists, Sarasota, Florida
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - START Midwest, Grand Rapids, Michigan
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - UH Seidman Cancer Center, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - NEXT Oncology, San Antonio, Texas
  - START Mountain, West Valley City, Utah